CLINICAL TRIAL: NCT06678984
Title: Treated Umbilical Vein Allograft (UVT) Versus Autologous Fascial Pubovaginal Sling in the Treatment of Female Stress Urinary Incontinence
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UVT-TBF2; 2024-A00352-45 (Other: IDRCB)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Stress Urinary Incontinence in Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated umbilical vein allograft (Experimental)
  Interventions: Procedure: with treated umbilical vein allograft
- Autologous Fascial Pubovaginal Sling (Active Comparator)
  Interventions: Procedure: with autologous fascial pubovaginal sling

INTERVENTIONS:
Procedure: with treated umbilical vein allograft — Surgical treatment of female stress urinary incontinence using a treated allogeneic umbilical vein sling
  Arms: Treated umbilical vein allograft
Procedure: with autologous fascial pubovaginal sling — Surgical treatment of female stress urinary incontinence using a autologous fascial pubovaginal sling
  Arms: Autologous Fascial Pubovaginal Sling

SUMMARY:
The goal of this clinical trial is to evaluate whether a treated umbilical vein allograft is effective in treating stress urinary incontinence in females. The researchers will compare the treated umbilical vein allograft with a sling made of autologous tissue. The main question the clinical trial aims to answer is:

- Is the treated umbilical vein allograft as effective as the sling made of autologous tissue for treating female stress urinary incontinence?

Participants will:

* Undergo surgical treatment with either the umbilical vein allograft or the sling made of autologous tissue on Day 0.
* Visit the hospital for a series of tests at 3 weeks, 3 months, 6 months, and 12 months after the surgical intervention.
* Record their bladder activity between each hospital visit.

DETAILED DESCRIPTION:
It is estimated that more than 9 million French people are affected by urinary incontinence, of which 1% are treated surgically. When medical management or rehabilitation fails, surgical treatment must be considered. Sling implantation is a commonly used surgical technique for treating stress urinary incontinence, as it reduces surgery time and morbidity, and can be performed under local anesthesia. However, the risk of complications associated with the use of synthetic materials is significant, contributing to a recent decline in the popularity of synthetic slings.

Given the high demand for incontinence treatments, autologous fascia sling surgeries are being proposed, despite requiring an additional surgical procedure and exposing patients to complications at the donor site of the graft.

The study product aims to address the need for a safer, equally effective implant that eliminates the need for autografting while maintaining standard surgical techniques.

The aim of this comparative study is to determine whether the efficacy of the treated umbilical vein allograft can justify its use as a substitute for the autologous fascial sling, thereby avoiding the complications associated with harvesting the autograft.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 85 years.
* Patients with stress urinary incontinence or mixed urinary incontinence with a predominant stress component.
* Patients with stress urinary incontinence due to cervico-urethral hypermobility or urethral hypermobility.
* Patients with urethral hypermobility confirmed by Ulmsten suburethral support maneuver.
* Urinary incontinence demonstrated by one-hour pad test.
* Patients with significant and persistent discomfort despite perineal rehabilitation.
* Patients able to understand the information concerning the study and having voluntarily dated and signed the informed consent form.
* Patients able and willing to comply with the requirements and instructions of the study.
* Patients who are members or the beneficiary of a national health insurance plan.

Exclusion Criteria:

* Pregnant or breastfeeding women or those not using effective contraception.
* Patients with a body mass index (BMI) ≥ 35 kg/m2.
* Patients with moderate stress urinary incontinence treated with physiotherapy and pelvic support exercises.
* Patients with voiding disorders or at risk of performing self-catheterization.
* Patients who have already undergone surgical treatment for urinary incontinence.
* Patients unable to perform the pad test or unwilling to perform it at each follow-up visit.
* Patients considered by the principal investigator to be poor candidates for surgical procedures and/or anesthesia due to their physical or mental state.
* Patients with current urinary tract infection, severe anemia, uncontrolled diabetes or other conditions contraindicating surgery.
* Patients with neurogenic bladder.
* Patients with a history of conditions, illnesses or surgical procedures that may confound the results of the urinary incontinence assessment, including but not limited to: pelvic organ prolapse (e.g., cystocele, rectocele), neurological disorders (e.g., multiple sclerosis, Parkinson's disease), recurrent urinary tract infections, recurrent bladder stones, interstitial cystitis, history of pelvic irradiation (external beam therapy or brachytherapy), current diagnosis of genitourinary malignancy.
* Patients deprived of liberty by a judicial or administrative decision.
* Patients incapable of discernment for rehabilitation, unable to follow up or give consent.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Difference between treatment groups in change from baseline to final 12-month postoperative visits in the amount of urinary leakage. | 12 months
  The amount of urinary leakage (grams) will be quantified by a one-hour pad test performed during patient visit at the hospital.
  One-hour pad test will be performed in the following way:
  * Subject puts on one standardized, pre-weighed pad without voiding.
  * 0-15 Minutes: Subject drinks 500 mL of sodium-free liquid in < 15 min while sitting or resting.
  * 15 - 45 Minutes: Subject walks for 30 minutes, including climbing one flight of stairs (up and down).
  * 45 - 60 Minutes: Subject performs the following activities: Standing up from sitting (10 times), Coughing vigorously (10 times), Running on the spot (1 min), Bending to pick up an object from the floor (5 times), Wash hands in running water (1 min).
  * The weight of the pad is measured to determine the amount of leakage.

SECONDARY OUTCOMES:
Difference between treatment groups in change from baseline to 3- and 6-month postoperative visits in the amount of urinary leakage. | 3 months, 6 months
  The amount of urinary leakage (grams) will be quantified by a one-hour pad test performed during patient visits at the hospital.
Difference between treatment groups in the proportion of subjects who achieved a reduction of more than 50% in the amount of urinary leakage between baseline and the 12-month visit. | 12 months
  The amount of urinary leakage (grams) will be quantified by a one-hour pad test performed during patient visit at the hospital.
Difference between treatment groups in change from baseline to final 12-month postoperative visits in the number of incontinence episodes and pads used daily. | 12 months
  The number of incontinence episodes and pads used daily will be determined from a voiding calendar carried out by the patient at home over a 3-day period.
Difference between treatment groups in changes between initial and postoperative visits in frequency, severity and impact on quality of life of patients' urinary incontinence, as measured by the ICIQ-UI-SF. | 3 months, 6 months, 12 months
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) assess frequency, severity and impact on quality of life (QoL) of patients' urinary incontinence symptoms. The result of the ICIQ-UI SF is a composite score ranging from 0 to 21, with higher scores indicating more severe incontinence.
Difference between treatment groups in changes between initial and postoperative visits in the distress caused by urinary incontinence symptoms, as measured by the UDI-6. | 3 months, 6 months, 12 months
  The Urogenital Distress Inventory (UDI-6) assess the distress caused by urinary incontinence symptoms. The UDI-6 total score ranges from 0 to 100, with higher scores indicating more distressing symptoms.
Difference between treatment groups in changes between initial and postoperative visits in the psychosocial impact of urinary incontinence in patients, as measured by the IIQ-7. | 3 months, 6 months, 12 months
  The Incontinence Impact Questionnaire (IIQ-7) assess the psychosocial impact of urinary incontinence in female patients. The IIQ-7 total score ranges from 0 to 100, with higher scores indicating a greater psychosocial impact of urinary incontinence on the patient.
Difference between treatment groups in changes between initial and postoperative visits in the patients' perceived symptom improvement, as measured by the PGI-I | 3 months, 6 months, 12 months
  Patients' perceived improvement in urinary incontinence symptoms will be assessed with the Patient Global Impression of Improvement (PGI-I). PGI-I measures improvement on a scale of 1 "very much better" to 7 "very much worse."
Difference between treatment groups in rates of specific complications | 3 weeks, 3 months, 6 months, 12 months
  Rate of specific complications, including skin reaction, delayed healing, urinary retention, injury to the bladder or other abdominal structures, severe and persistent pain will be evaluated during each patient's post-operative visits to the hospital.

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Hôpital Estaing, CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hôpital Michalon, CHU de Grenoble Alpes, La Tronche
  - Hôtel-Dieu, CHU de Nantes, Nantes
  - Hôpital de la Pitié-Salpêtrière, Assistance Publique des Hôpitaux de Paris, Paris
  - Hôpital Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite
  - Hôpital Charles-Nicolle, CHU de Rouen, Rouen
  - Nouvel hôpital civil, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital Rangueil, CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No